CLINICAL TRIAL: NCT00545415
Title: The Effect of Fruit and Fruit Juice on Plasma Total Antioxidant Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Aalt Bast, Prof. Dr., Maastricht University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MEC-07-3-043
Record Dates: First submitted 2007-10-11; First posted 2007-10-17 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2009-07

CONDITIONS: Healthy
Keywords: fruit; antioxidant; Healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Dietary Supplement: Order 1
- 2 (Experimental)
  Interventions: Dietary Supplement: Order 2
- 3 (Experimental)
  Interventions: Dietary Supplement: Order 3
- 4 (Experimental)
  Interventions: Dietary Supplement: Order 4
- 5 (Experimental)
  Interventions: Dietary Supplement: Order 5
- 6 (Experimental)
  Interventions: Dietary Supplement: Order 6

INTERVENTIONS:
Dietary Supplement: Order 1 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 1
Dietary Supplement: Order 2 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 2
Dietary Supplement: Order 3 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 3
Dietary Supplement: Order 4 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 4
Dietary Supplement: Order 5 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 5
Dietary Supplement: Order 6 — Supplement is fruit, fruit salad and fruit drink in different order. Fruit (two apples) Fruit salad, 400g (consist of apple, banana, orange, mandarin, pear, strawberry, grape, kiwi and melon) in amount relative to the popularity of the fruits consumed in the Netherlands.
  Fruit drink (fruit2day, strawberry/orange, 200ml) Each supplement is taken once, with one week wash out.
  Arms: 6

SUMMARY:
The aim of the study is to compare the effect of consumption of a fruit beverage on plasma antioxidant capacity with that of the consumption of fruit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* body mass index between 20-25

Exclusion Criteria:

* use of any medication
* smoking
* consumption of 3 or more glasses of alcohol per day
* involved in top sport

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The total plasma antioxidant capacity after intake of three different kinds of fruit(beverage) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Netherlands